CLINICAL TRIAL: NCT02420080
Title: A Multicenter Non-Interventional Study to Obtain Retrospective Data for Subjects Previously Diagnosed With Adenovirus Infection to Serve as Matched Historical Controls for Study CMX001-304
Brief Title: A Multicenter Study to Obtain Retrospective Data for Subjects Previously Diagnosed With Adenovirus Infection to Serve as Matched Historical Controls for Study CMX001-304
Status: Terminated | Type: Observational
Why Stopped: Study was terminated early due to results from previous CMX study
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CMX001-305
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Adenovirus
MeSH Terms: conditions — Adenoviridae Infections | interventions — brincidofovir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: The primary endpoint for subjects in Cohort A is time to progression of AdV disease through Week 24 post initial AdV diagnosis, with progression of AdV disease defined as time to the following outcomes:
  Clinical progression to probable or definitive disseminated AdV disease Death
  Interventions: Drug: Brincidofovir
- Cohort B: The primary endpoint for subjects in Cohort B is time to all-cause mortality through Week 36 post diagnosis of disseminated AdV disease
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — Rates of adenovirus progression and mortality in subjects with adenovirus infection and/or disease. Sites participating in the CMX001-304 study will be asked to participate in the CMX001-305 study retrospective data collection study.
  Other Names: CMX001

SUMMARY:
The objective is data collection to determine background rates of adenovirus (AdV) progression and mortality in subjects with Adenovirus (AdV) infection and/or disease.

DETAILED DESCRIPTION:
The objective of this retrospective data collection is to determine background rates of adenovirus (AdV) progression and mortality in subjects with Adenovirus (AdV) infection and/or disease.

ELIGIBILITY:
Inclusion Criteria:

* Matched-control cases must be recruited from sites participating in the CMX001-304 study and meet all of the following criteria, as applicable, to be eligible for data abstraction in this non-interventional retrospective study:
* Age at time of transplant: ≥ 2 months
* Eligible matched-control subjects must meet the disease conditions of one or both of the two cohorts listed below on or after Jan 1, 2004 and prior to Mar 12, 2014. If subjects had more than one study-qualifying episode of these disease conditions on or after Jan 1, 2004 and prior to Mar 12, 2014, only the most recent qualifying episode should be included:
* Cohort A: allogeneic hematopoietic cell transplantation (HCT) recipients who were at risk of progression to disseminated AdV disease, defined as documented evidence of 1) asymptomatic AdV viremia ≥ 1,000 copies/mL, increasing, OR 2) localized AdV infection
* Cohort B: allogeneic HCT recipients with disseminated AdV disease

Exclusion Criteria:

* Prior use of BCV

Ages: 2 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: allogeneic hematopoietic cell transplant (HCT) recipients who were at risk of progression to disseminated AdV disease. Allogeneic hematopoietic cell transplant recipients with disseminated AdV disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cohort A (Time to progression of AdV disease through Week 36) | 36 weeks
  Time to progression of AdV disease through Week 36 post initial AdV diagnosis, with progression of AdV disease defined as time to the occurrence of either clinical progression to probable or definitive disseminated AdV disease or Death.

SECONDARY OUTCOMES:
Cohort B (Time to all-cause mortality through Week 36) | 36 weeks
  Time to all-cause mortality through Week 36 post diagnosis of disseminated AdV disease

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Childrens National Health System, Washinton, District of Columbia
  - Emory University, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hosital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Judes Children's Research Hospital, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Utah Cancer Specialist LDS Hospital, Salt Lake City, Utah
  - University of Washington_Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin